CLINICAL TRIAL: NCT01230528
Title: Childhood Reactive Thrombocytosis (RT)
Brief Title: Childhood Reactive Thrombocytosis
Acronym: RT
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Jinn-Li Wang, Department of Pediatrics, WanFang Hospital
Other Study IDs: WFH-PED 002 Version.2/990603
Record Dates: First submitted 2010-10-27; First posted 2010-10-29 (Estimated); Last update posted 2010-10-29 (Estimated); Status verified 2010-10

CONDITIONS: Reactive Thromobocytosis in Children

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Reactive thrombocytosis (RT) in pediatric patients is common, but usually without symptoms. The incidence of RT is different depending on age. Mostly, we reasoned that RT is a phenomenon, nevertheless the diagnostic value of RT is little known. Therefore, the aim of this study was to determine the association of RT and clinical or laboratory characteristics in pediatric diseases.

ELIGIBILITY:
Inclusion Criteria:

* The platelet counts more than 500x109/l and age less than 18 years old.

Exclusion Criteria:

* repeated hospitalization ( more than 2 times)

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The investigators will enroll all pediatric hospitalized patients with platelet counts more than (500x109/l) at complete blood counts examination.The association of reactive thrombocytosis and clinical manifestation will be analyzed.
Sampling Method: Probability Sample
Dates: Start 2009-07; Primary Completion 2010-01 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jinn-Li Wang, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University-WanFang Hospital, Taipei, Taiwan